CLINICAL TRIAL: NCT02554591
Title: Retrospective Analysis of Genomic Landscape of ALK Positive NSCLC Prior to Ceritinib, and at Disease Progression Following Ceritinib
Brief Title: Genomic Landscape of Ceritinib
Status: Terminated | Type: Observational
Why Stopped: Changes in treatment plans affecting drug therapy choices
Sponsor: Washington University School of Medicine (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 201509030
Record Dates: First submitted 2015-09-08; First posted 2015-09-18 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Non-small Lung Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators propose to conduct a retrospective study of single agent ceritinib in patients with previously untreated anaplastic lymphoma kinase (ALK) rearranged adenocarcinoma of the lung with the sole purpose of characterizing the genomic landscape before ceritinib and at the time of disease progression.

DETAILED DESCRIPTION:
Further improvements in therapy can only be achieved with a better understanding of the genomic landscape of ALK rearranged non-small cell lung cancer (NSCLC), specifically at the time of disease progression following treatment with ALK inhibitors. Recently, secondary ALK mutations, L1196M and G1269A have been described in patients with acquired resistance to crizotinib. A small subset of ALK positive lung cancer patients who progressed after treatment with ceritinib had tumors available for molecular analysis. Secondary mutations found included G1202R, F1174C, and F1174V. While this is interesting, an unbiased genomic study (exome or whole genome sequencing) using massively parallel sequencing at the time of disease progression is critical to fully understand the clonal evolution and the molecular mechanisms underpinning treatment resistance. To the best of the investigators' knowledge, such a study has not yet been reported.

The investigators believe the time is ripe now to comprehensively characterize genomic alterations using massively parallel sequencing technology of ALK driven adenocarcinoma of the lung to fully understand the clonal heterogeneity before therapy and fully understand the clonal evolution and the molecular mechanisms underpinning treatment resistance. A better understanding of genomic alterations through an unbiased comprehensive approach likely would lead to rationally designed therapy to augment response to ALK inhibitors.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of metastatic stage IIIB/IV lung adenocarcinoma.
* Presence of known ALK gene rearrangement.
* Consented to HRPO# 201305031 ("Tissue and Blood Acquisition for Genomic Analysis and Collection of Health Information from Patients with Thoracic Malignancies, Suspected Thoracic Malignancies, or Mesothelioma") with an existing specimen prior to initiation of treatment with ceritinib.
* At least 18 years of age.
* Received treatment with standard of care ceritinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the Washington University School of Medicine and Barnes-Jewish healthcare system who previously consented to study HRPO (Human Research Protection Office)# 201305031 ("Tissue and Blood Acquisition for Genomic Analysis and Collection of Health Information from Patients with Thoracic Malignancies, Suspected Thoracic Malignancies, or Mesothelioma").
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Genetic changes associated with disease progression following treatment with ceritinib | Estimated to be 1 year
  * The investigators will compare tumor sequencing prior to ceritinib treatment to the time of disease progression to see if the genetic sequencing changed between pre-treatment and progression.
  * The investigators plan to conduct exome and transcriptome sequencing of tumor before therapy with certitinib and at the time of relapse. In addition, exome sequencing of peripheral blood DNA will be done (for germline). Given the complexities of genomic analyses of paired samples in the face of limited data, the investigators will not be able to do any formal power calculations in this feasibility study.
  * Disease progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.

SECONDARY OUTCOMES:
Types of mutations in signaling kinases associated with therapeutic response | Estimated to be 1 year
  * Investigators will look at tumor tissue associated with a therapeutic response and compare with tumor tissue associated with disease progression and see if there are any mutation differences.
  * Therapeutic Response
    * Complete response is disappearance of all target lesions and non-target lesions.
      * Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Allelic ratio of wild type ALT to ALK gene rearrangement (roughly corrected for intrinsic difference in tumor cellularity) with duration of response | Estimated to be 1 year
  * A variant is considered to have mutant biased expression if the variant is expressed and the variant allele frequency is greater than 20% higher in the RNA-seq data compared to the exome sequencing data. A variant is considered to have wild type biased expression if the gene is expressed, the region of the variant is covered at 5X or greater depth, and the VAF is at least 20% lower in the RNA-seq data compared to the exome sequencing data.
  * Duration of response is the duration of overall response is measured from the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu